CLINICAL TRIAL: NCT06288529
Title: PROTECTIVE EFFECT OF SGLT2 INHIBITORS ON POST-CONTRAST MEDIUM INDUCED ACUTE KIDNEY INJURY IN DIABETIC AND CKD PATIENTS
Brief Title: EFFECT SGLT2 INHIBITORS ON CONTRAST MEDIUM INDUCED ACUTE KIDNEY INJURY
Status: Completed | Type: Observational
Sponsor: University of Health Sciences Balikesir Hospital Eduation and Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Kidney Diseases; Type2diabetes
Keywords: Sodium-glucose co-transporter inhibitor; post-contrast acute kidney injury; contrast media; diabetes mellitus; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients with type 2 diabetes mellitus using SGLT2 inhibitor
- Patients with type 2 diabetes mellitus not using SGLT2 inhibitor
- Patients with chronic kidney disease mellitus using SGLT2 inhibitor
- Patients with chronic kidney disease mellitus not using SGLT2 inhibitor

SUMMARY:
Chronic kidney disease and type 2 diabetes mellitus patients are with in high-risk patients in coronary arterial diseases and increasing number of coronary angiography and coronary interventional procedures have been performed in these population. As well as the risk factors have been identified by many studies preventive measures are lacking.

In our study we found that SGLT2 inhibitors are beneficial in terms of reducing contrast media induced acute kidney injury in both diabetic and CKD patients.This is one of the leading studies in the literature pointing that SGLT2 inhibitors may have a potentially beneficial role in reducing or preventing the development of PC-AKI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent coronary artery imaging or percutaneous coronary intervention procedures using contrast media
* Patient ages were between 18 and 75 years
* Estimated glomerular filtration rates (eGFRs) between 25 and 115

Exclusion Criteria:

* Patients with acute myocardial infarction, acute renal injury, history of kidney transplantation, severe heart failure (HF, New York Heart Association IV), malignancy, also patients who received other PC-AKI preventive medications like as N-acetylcysteine, sodium bicarbonate, or incomplete medical records were excluded from the analyses.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Total of 975 patients are palanned to be included in our study who underwent coronary artery imaging or percutaneous coronary intervention procedures using CM in three tertiary hospitals. Patient ages between 18 and 75 years and estimated glomerular filtration rates (eGFRs) between 25 and 115 mL/(min•1.73 m2) are palanned to be included in our analyses.
Sampling Method: Non-Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Development of post-contrast acute kidney injury | Within 48-72 hours following intravenous contrast medium administration.
  The impairment of renal function which is measured as either a 25% rise in serum creatinine level from baseline or an increase of 0.5 mg/dL (44 µmol/L) in absolute serum creatinine level.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Balikesir Education and Research Hospital, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided